CLINICAL TRIAL: NCT03014375
Title: An Open-label Study in Healthy Male Subjects to Assess the Absorption, Distribution, Metabolism and Excretion of [14C]-Labeled BIA 5-453 and Metabolites Following a Single-dose Oral Administration
Brief Title: Absorption, Distribution, Metabolism and Excretion of [14C]- Labeled BIA 5-453 and Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-5453-103
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension; Congestive Heart Failure
MeSH Terms: conditions — Hypertension; Heart Failure | interventions — etamicastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etamicastat (Experimental): Single administration. 100 μCi/ 3.7 MBq 14C labeled BIA 5-453 50 mg, hard gelatina capsules
  Interventions: Drug: BIA-5-453

INTERVENTIONS:
Drug: BIA-5-453 — Each subject will receive a single oral dose of 100 μCi/ 3.7 MBq 14C labeled BIA 5-453 (600 mg).

SUMMARY:
The purpose of this study is to:

To determine the rate and routes of excretion of BIA 5-453 and the mass balance in urine and faeces

DETAILED DESCRIPTION:
Monocentre, open, non-placebo-controlled, single-group, single-dose study Safety measurements (12-lead ECG, vital signs, blood chemistry and haematology) will be conducted before and after the study, adverse events will be monitored throughout the study.

Subjects should be hospitalized the day before the administration until 264 hours thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian male subjects, 40-55 years of age.
* Sitting blood pressure and pulse rate within a clinically acceptable range for the purposes of the study, i.e.: BP: 100 160 mmHg systolic, 50 95 mmHg diastolic and pulse rate: 50 100 bpm. Blood pressure and pulse will be measured after 3 minutes resting in a sitting position.
* Subject body mass index must be between 18 and 28 kg/m2
* Normal 12-lead ECG
* Ability to communicate well with the investigator and comply with the requirements of the entire study.
* The subject has given his written informed consent to participate in the study.

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug.
* Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
* History of alcohol or drug abuse in the last 5 years.
* Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
* Need of any prescription medication within 14 days prior to the administration of the drug and/or nonprescription medication within 7 days prior to the administration of the drug.
* Participation in other clinical trials during the previous month in which an investigational drug or a commercially available drug was tested.
* Loss of 500 mL blood or more during the 3 month period before the study, e.g., as a donor.
* Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e., impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhoea or conditions associated with total or partial obstruction of the urinary tract.
* Symptoms of a significant somatic or mental illness in the 4 week period preceding drug administration.
* History of hepatitis B and / or C and / or positive serology results which indicate the presence of hepatitis B and / or C.
* Positive results from the HIV serology.
* Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening evaluation, however, liver parameters (SGPT, SGOT) values must be within the normal range.
* Positive results of the drug screening.
* Known hypersensitivity to BIA 5-453.
* Heavy smokers, i.e., more than 10 cigarettes per day
* Exposure to artificial ionizing radiation in the last 12 months (e.g., x-ray investigation)
* Subject who had more than 4 flights (with more than 2 hours flight time) within the last year prior to the administration of the drug

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
urinary excretion of BIA 5-453 associated radioactivity | pre-dose, then it was collected from 0-4, 4-8, 8-24, 24-48, 48-72, 72-120, 120-168, 168-216, and 216-264 hours post-dose.
  following a single 600 mg oral dose labeled with 98 μCi of [14C]
faecal excretion of BIA 5-453 associated radioactivity | following a single 600 mg oral dose labeled with 98 μCi of [14C]
  baseline period. Following dose, each faeces sample was collected during the 264 hours post-dose period.
amount of BIA 5-453 associated radioactivity present in the expired air | baseline, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h 6h, 8h, 12h and 24h post-dose
  following a single 600 mg oral dose labeled with 98 μCi of [14C]

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Pharma Contract Ltd., Allschwil, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided